CLINICAL TRIAL: NCT05675410
Title: A Randomized Phase 3 Interim Response Adapted Trial Comparing Standard Therapy With Immuno-oncology Therapy for Children and Adults With Newly Diagnosed Stage I and II Classic Hodgkin Lymphoma
Brief Title: A Study to Compare Standard Therapy to Treat Hodgkin Lymphoma to the Use of Two Drugs, Brentuximab Vedotin and Nivolumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-10845; NCI-2022-10845 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AHOD2131 (Other: Children's Oncology Group); AHOD2131 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-01-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Lugano Classification Limited Stage Hodgkin Lymphoma AJCC v8
MeSH Terms: interventions — Specimen Handling; Bleomycin; Brentuximab Vedotin; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; etoposide phosphate; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Nivolumab; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; Procarbazine; Vinblastine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm A (ABVD) (Active Comparator): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive ABVD IV for an additional 2 cycles on study. Each cycle lasts 28 days and ABVD is administered on days 1 and 15 of each cycle in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate
- Arm B (ABVD, brentuximab vedotin, nivolumab) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30 minutes once during each treatment cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate
- Arm C (ABVD, eBEACOPP or eBPDac, ISRT) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Etoposide Phosphate; Other: Fludeoxyglucose F-18; Radiation: Involved-site Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Drug: Procarbazine Hydrochloride; Other: Questionnaire Administration; Drug: Vinblastine Sulfate; Drug: Vincristine Sulfate
- Arm D (ABVD, brentuximab vedotin, nivolumab, ISRT) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive brentuximab vedotin IV and nivolumab IV as in arm B followed by ISRT. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Radiation: Involved-site Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate
- Arm E (ABVD, AVD) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive AVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, vinblastine IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate
- Arm F (ABVD, brentuximab vedotin, nivolumab) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive treatment as in arm B. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate
- Arm G (ABVD, eBEACOPP or eBPDac, ISRT) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive treatment and imaging, and may undergo blood sample collection as in arm C.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Etoposide Phosphate; Other: Fludeoxyglucose F-18; Radiation: Involved-site Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Drug: Procarbazine Hydrochloride; Other: Questionnaire Administration; Drug: Vinblastine Sulfate; Drug: Vincristine Sulfate
- Arm H (ABVD, brentuximab vedotin, nivolumab, ISRT) (Experimental): Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or MRI and are identified as RER or SER. Patients then receive treatment and imaging, and may undergo blood sample collection as in arm D.
  Interventions: Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Fludeoxyglucose F-18; Radiation: Involved-site Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Vinblastine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Bleomycin Sulfate — Given IV
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Bleomycini Sulfas; Blexane; Oil Bleo
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
  Arms: Arm B (ABVD, brentuximab vedotin, nivolumab); Arm D (ABVD, brentuximab vedotin, nivolumab, ISRT); Arm F (ABVD, brentuximab vedotin, nivolumab); Arm H (ABVD, brentuximab vedotin, nivolumab, ISRT)
Procedure: Computed Tomography — Undergo CT and/or PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Other: Fludeoxyglucose F-18 — Undergo FDG-PET
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Involved-site Radiation Therapy — Undergo ISRT
  Other Names: ISRT
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm D (ABVD, brentuximab vedotin, nivolumab, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT); Arm H (ABVD, brentuximab vedotin, nivolumab, ISRT)
Procedure: Magnetic Resonance Imaging — Undergo MRI and/or PET-MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm B (ABVD, brentuximab vedotin, nivolumab); Arm D (ABVD, brentuximab vedotin, nivolumab, ISRT); Arm F (ABVD, brentuximab vedotin, nivolumab); Arm H (ABVD, brentuximab vedotin, nivolumab, ISRT)
Procedure: Positron Emission Tomography — Undergo FDG-PET, PET, PET-CT, and/or PET-MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisolone — Given PO
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Drug: Procarbazine Hydrochloride — Given PO
  Other Names: Benzamide, N-(1-methylethyl)-4-[(2-methylhydrazino) methyl]-, monohydrochloride (9CI); Ibenzmethyzine hydrochloride; Matulane; MIH hydrochloride; Natulan; Natulanar; Natunalar; NCI C01810; NCI-C01810; NCIC01810; p-(N'-methylhydrazinomethyl)-N-isopropylbenzamide hydrochloride; p-Toluamide, N-isopropyl-.alpha.-(2-methylhydrazino)-, monohydrochloride (8CI); PCB; PCB Hydrochloride; PCZ; Ro 4 6467/1; Ro 4-6467/1
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)
Other: Questionnaire Administration — Ancillary studies
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm C (ABVD, eBEACOPP or eBPDac, ISRT); Arm G (ABVD, eBEACOPP or eBPDac, ISRT)

SUMMARY:
This phase III trial compares the effect of adding immunotherapy (brentuximab vedotin and nivolumab) to standard treatment (chemotherapy with or without radiation) to the standard treatment alone in improving survival in patients with stage I and II classical Hodgkin lymphoma. Brentuximab vedotin is in a class of medications called antibody-drug conjugates. It is made of a monoclonal antibody called brentuximab that is linked to a cytotoxic agent called vedotin. Brentuximab attaches to CD30 positive lymphoma cells in a targeted way and delivers vedotin to kill them. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs such as doxorubicin hydrochloride, bleomycin sulfate, vinblastine sulfate, dacarbazine, and procarbazine hydrochloride work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill cancer cells. It may also lower the body's immune response. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Adding immunotherapy to the standard treatment of chemotherapy with or without radiation may increase survival and/or fewer short-term or long-term side effects in patients with classical Hodgkin lymphoma compared to the standard treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) of a standard chemotherapy approach versus an immunotherapy (IO) approach (brentuximab vedotin and nivolumab) in patients with newly diagnosed early stage classic Hodgkin lymphoma (cHL) who have a rapid early response (RER) as determined by position emission tomography post cycle 2 (PET2) after 2 cycles of doxorubicin, bleomycin, vinblastine, dacarbazine (ABVD) chemotherapy.

II. To compare the PFS of a standard chemotherapy approach versus an IO therapy approach (brentuximab vedotin and nivolumab) plus involved site radiation therapy (ISRT) in patients with newly diagnosed early stage cHL who have a slow early response (SER) as determined by PET2 after 2 cycles of ABVD chemotherapy.

SECONDARY OBJECTIVES:

I. To demonstrate non-inferiority of overall survival (OS) at 12 years of IO therapy versus standard therapy in early stage cHL patients who have a RER as determined by PET2 after 2 cycles of doxorubicin, bleomycin, vinblastine, dacarbazine (ABVD) chemotherapy.

II. To evaluate the overall survival (OS) at 12 years of IO therapy versus standard therapy in early stage cHL patients who have a SER as determined by PET2 after 2 cycles of doxorubicin, bleomycin, vinblastine, dacarbazine (ABVD) chemotherapy.

III. To demonstrate non-inferiority of overall survival (OS) at 12 years of IO therapy versus standard therapy in early stage cHL patients.

IV. To evaluate in patients with newly diagnosed early stage cHL the PFS of a standard chemotherapy approach versus an IO therapy approach (brentuximab vedotin and nivolumab) in the overall cohort, in the favorable risk cohort, and in the unfavorable risk cohort.

V. To evaluate the event-free survival (EFS) at 12 years of patients undergoing standard chemotherapy versus an IO therapy approach (brentuximab vedotin and nivolumab).

VI. To compare the physician-reported treatment-related adverse event (AE) rates between a standard chemotherapy approach and an IO therapy approach (brentuximab vedotin and nivolumab) in patients with newly diagnosed early stage cHL.

VII. To compare patient-reported adverse events using pediatric and adult versions of Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), stratified by age groups, therapeutic arms, and receipt of radiation therapy (RT) over time.

VIII. To evaluate changes in patient-reported fatigue, cognitive functioning, and health-related quality of life (HRQoL), e.g., emotional, physical, and role functioning, by treatment arm, using validated adult and pediatric measurement systems.

IX. To evaluate self-reported late morbidities (e.g., cardiovascular, pulmonary and endocrine) over time for children, adolescents and adults undergoing standard chemotherapy versus an IO therapy approach (brentuximab vedotin and nivolumab) with and without RT using measures from the St. Jude Lifetime Cohort Study (SJLIFE).

X. To evaluate fludeoxyglucose F-18 (FDG)-position emission tomography (PET) measurements of metabolic tumor burden (MTV and total lesion glycolysis [TLG]) at PET at baseline (PET1) as a predictive marker of PFS.

XI. To evaluate the associations between race/ethnicity and key outcomes including early response to therapy, PFS and OS.

EXPLORATORY OBJECTIVES:

I. To evaluate the PFS of a standard chemotherapy approach versus an IO therapy approach (brentuximab vedotin and nivolumab) in patients with newly diagnosed early stage cHL across different age groups (ages 5-11 years, 12-21 years, 22-39 years, 40-60 years).

II. To bank specimens for future correlative studies. III. To assess concordance and discordance of rapid central review and local institutional review of FDG PET 5-point score (5-PS; previously referred to as Deauville score) at baseline PET1, interim PET2 and end of systemic therapy PET-end of systemic therapy (EST) SER.

IV. To assess the association between PFS and the quantitative FDG-PET/computed tomography (CT) parameters (PET MTV, TLG, delta-standardized uptake value [SUV] and PET SUV-based quantitative surrogates [qPET] of visual qualitative 5-PS) on measurements by automated measurements using convolutional neural networks (CNNs) through artificial-intelligence (AI) machine learning in the entire population.

V. To assess the agreement between quantitative FDG-PET/CT parameters obtained using AI and those based on measurements by a trained imaging physician.

VI. To compare patient-reported adverse events (via pediatric [Ped]-PRO-CTCAE and PRO-CTCAE) to provider adverse event reporting.

VII. To evaluate the association between self-reported race/ethnicity and social determinants of health.

VIII. To evaluate the associations between race/ethnicity and post-progression/post-relapse overall survival.

IX. To evaluate the completion rates of PRO and health-related quality of life (HRQoL) contact forms at 1 year off treatment for the first 450 eligible patients.

X. To collect contact information from participants for future re-contact.

OUTLINE: Patients are stratified by risk status (favorable versus unfavorable) and then all patients receive the ABVD regimen (doxorubicin hydrochloride intravenously [IV] over 3-15 minutes, bleomycin sulfate IV over at least 10 minutes, vinblastine sulfate IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo FDG-PET/CT or magnetic resonance imaging (MRI) and are identified as RER or SER.

Patients with a favorable risk status and RER are randomized to Arm A or Arm B. Patients with a favorable risk status and SER are randomized to Arm C or Arm D. Patients with an unfavorable risk status and RER are randomized to Arm E or Arm F. Patients with an unfavorable risk status and SER are randomized to Arm G or Arm H.

ARM A (RER, FAVORABLE): Patients receive ABVD IV for an additional 2 cycles on study. Each cycle lasts 28 days and ABVD is administered on days 1 and 15 of each cycle in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM B (RER, FAVORABLE): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30 minutes once during each treatment cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM C (SER, FAVORABLE): Patients receive either the eBEACOPP regimen (doxorubicin hydrochloride IV over 3-15 minutes on day 1, cyclophosphamide IV over 30-60 minutes on day 1, etoposide or etoposide phosphate IV over 2-4 hours on days 1-3, prednisone or prednisolone orally [PO] twice daily [BID] on days 1-14, procarbazine hydrochloride PO on days 1-7, bleomycin sulfate IV over at least 10 minutes on day 8, and vincristine sulfate IV on day 8 of each cycle) or the eBPDac regimen (doxorubicin hydrochloride IV 3-15 minutes on day 1, cyclophosphamide IV 30-60 minutes on day 1, etoposide or etoposide phosphate IV over 2-4 hours on days 1-3, prednisone or prednisolone PO BID on days 1-14, dacarbazine IV over 15-60 minutes on days 2 & 3, bleomycin sulfate IV over at least 10 minutes on day 4, 5, 6, 7, or 8, vincristine sulfate IV on day 4, 5, 6, 7, or 8 of each cycle). Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Subsequently, patients undergo ISRT. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM D (SER, FAVORABLE): Patients receive brentuximab vedotin IV and nivolumab IV as in arm B followed by ISRT. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM E (RER, UNFAVORABLE): Patients receive AVD regimen (doxorubicin hydrochloride IV over 3-15 minutes, vinblastine IV, and dacarbazine IV over 15-60 minutes) on days 1 and 15 of each treatment cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM F (RER, UNFAVORABLE): Patients receive treatment as in arm B. Patients also undergo FDG-PET, PET, PET-CT, PET-MRI, CT, and/or MRI throughout the trial. Patients may also undergo blood sample collection on trial.

ARM G (SER, UNFAVORABLE): Patients receive treatment and imaging, and may undergo blood sample collection as in arm C.

ARM H (SER, UNFAVORABLE): Patients receive treatment and imaging, and may undergo blood sample collection as in arm D.

After completion of study treatment, patients are followed up every 3 months for the first year, then every 6 months for the second and third year, then annually until 12 years from date of registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 5 to 60 years of age at the time of enrollment
* Patients with newly diagnosed untreated histologically confirmed classic Hodgkin lymphoma (cHL) (nodular sclerosis, mixed cellularity, lymphocyte-rich, or lymphocyte-depleted, or not otherwise specified [NOS]) with stage I or II disease
* Patients must have bidimensionally measurable disease (at least one lesion with longest diameter >= 1.5 cm)
* Patients must have a whole body or limited whole body PET scan performed within 42 days prior to enrollment. PET-CT is strongly preferred. PET-MRI allowed if intravenous contrast enhanced CT is also obtained
* Pediatric patients (age 5-17 years) with known or suspected mediastinal disease must have an upright posteroanterior (PA) chest X-ray (CXR) for assessment of bulky mediastinal disease.

  * Note: Pediatric patients who have received both a CT chest and upright PA CXR may meet the definition of bulk through either modality.
* Patients >= 18 years must have a performance status corresponding to Zubrod scores of 0, 1 or 2
* Patients =< 17 years of age must have a Lansky performance score of >= 50
* Pediatric patients (age 5-17 years): A serum creatinine based on age/sex as follows (within 28 days prior to enrollment):

  * 2 to < 6 years (age): 0.8 mg/dL (male), 0.8 mg/dL (female)
  * 6 to < 10 years (age): 1 mg/dL (male), 1 mg/dL (female)
  * 10 to < 13 years (age): 1.2 mg/dL (male), 1.2 mg/dL (female)
  * 13 to < 16 years (age): 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years (age): 1.7 mg/dL (male), 1.4 mg/dL (female) OR a 24 hour urine creatinine clearance >= 50 mL/min/1.73 m^2 (within 28 days prior to enrollment) OR a glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (within 28 days prior to enrollment). GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
  * Note: Estimated GFR (eGFR) from serum or plasma creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* For adult patients (age 18 years or older) (within 28 days prior to enrollment): Creatinine clearance >= 30 mL/min, as estimated by the Cockcroft and Gault formula or a 24-hour urine collection. The creatinine value used in the calculation must have been obtained within 28 days prior to registration. Estimated creatinine clearance is based on actual body weight
* Total bilirubin =< 2 x upper limit of normal (ULN) (within 28 days prior to enrollment)

  * Unless due to Gilbert's disease, lymphomatous involvement of liver or vanishing bile duct syndrome
* Aspartate aminotransferase (AST) =< 3 x ULN (within 28 days prior to enrollment)

  * Unless due to Gilbert's disease, lymphomatous involvement of liver or vanishing bile duct syndrome
* Alanine aminotransferase (ALT) =< 3 x ULN (within 28 days prior to enrollment)

  * Unless due to Gilbert's disease, lymphomatous involvement of liver or vanishing bile duct syndrome
* Shortening fraction of >= 27% by echocardiogram (ECHO), multigated acquisition scan (MUGA), or functional cardiac imaging scan (within 28 days prior to enrollment) or ejection fraction of >= 50% by radionuclide angiogram, ECHO, MUGA, or cardiac imaging scan (within 28 days prior to enrollment)
* Diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% of predicted value as corrected for hemoglobin by pulmonary function test (PFT) (within 28 days prior to enrollment). If unable to obtain PFTs, the criterion is: a pulse oximetry reading of > 92% on room air
* Known human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

Exclusion Criteria:

* Patients with nodular lymphocyte predominant Hodgkin lymphoma
* Patients with a history of active interstitial pneumonitis or interstitial lung disease
* Patients with a diagnosis of inherited or acquired immunodeficiency that is poorly controlled or requiring active medications, such as primary immunodeficiency syndromes or organ transplant recipients
* Patients with any known uncontrolled intercurrent illness that would jeopardize the patient's safety such as infection, autoimmune conditions, cardiac arrhythmias, angina pectoris, and gastrointestinal disorders affecting swallowing and/or absorption of pills
* Patients with a condition requiring systemic treatment with either corticosteroids (defined as equivalent to > 10 mg daily predniSONE for patients >= 18 years or > 0.5 mg/kg [up to 10 mg/day] for patients < 18 years) or other immunosuppressive medications within 14 days prior to enrollment

  * Note: Replacement therapy such as thyroxine, insulin, or physiologic corticosteroid for adrenal or pituitary insufficiency is not considered a form of systemic treatment. Inhaled or topical steroids, and adrenal replacement doses (=< 10 mg daily for patients >= 18 years or =< 0.5 mg/kg [up to 10 mg/day] predniSONE equivalents) are permitted in the absence of active autoimmune disease
  * Note: Steroid use for the control of Hodgkin lymphoma symptoms is allowable, but must be discontinued by cycle 1, day 1
  * Short term use of corticosteroids for premedication or treatment of an allergy or hypersensitivity is considered an acceptable use of corticosteroids.
* Patients with peripheral neuropathy > grade 1 at the time of enrollment or patients with known Charcot-Marie-Tooth syndrome
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Administration of prior chemotherapy, radiation, or antibody-based treatment for cHL
* Prior solid organ transplant
* Prior allogeneic stem cell transplantation
* Live vaccine within 30 days prior to planned day 1 of protocol therapy (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, bacillus Calmette Guerin [BCG], oral polio vaccine, and oral typhoid). Administration of messenger ribonucleic acid (mRNA) vaccines are permitted
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test within 28 days prior to enrollment is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants starting with the first dose of study therapy and for at least 6 months after the last treatment
* Sexually active patients of reproductive potential who have not agreed to use a highly effective contraceptive method for the duration of their study drug therapy. Following therapy, patients will be advised to use contraception as per institutional practice or as listed below for investigational agents, whichever is longer

  * Men and women of childbearing potential (WOCBP) must use effective contraception during the study and for 2 months for WOCBP and 4 months for men, after last dose of brentuximab vedotin
  * WOCBP must continue contraception for a period of at least 5 months after the last dose of nivolumab
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1875 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2031-04-28 (Estimated); Study Completion 2031-04-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in rapid early responder (RER) patients | From the time of randomization to the earliest time of disease relapse, progression, or death due to any cause, assessed up to 3 years after the randomization of the last patient or when reaching 124 events, whichever comes first
  Will compare the PFS of RER patients randomized to immunotherapy (IO) therapy (brentuximab vedotin-nivolumab) against those randomized to standard therapy. PFS curves will be estimated separately by arm using Kaplan Meier methodology, and the test will be a 1-sided log-rank test between the (pooled) IO and standard arms, stratified according to the stratification factors at randomization and including all eligible and evaluable randomized patients.
PFS in slow-early responder (SER) patients | From the time of randomization to the earliest time of disease relapse, progression, or death due to any cause, assessed up to 3 years after the randomization of the last patient or when reaching 71 events, whichever comes first
  Will compare PFS among SER patients randomized to IO therapy and involved-site radiation therapy against arms containing standard therapy. PFS curves will be estimated separately by arm using Kaplan Meier methodology, and the test will be a 1-sided log-rank test between the (pooled) IO and standard arms, stratified according to the stratification factors at randomization and including all eligible and evaluable randomized patients.

SECONDARY OUTCOMES:
Overall survival (OS) in RER patients | Time from randomization to death due to any cause, assessed up to 12 years after the last enrollment
  The non-inferiority of IO therapy to standard therapy will be tested in the randomized and eligible RER cohort using a confidence interval approach performed 12 years after the last patient not lost to follow-up has reached more than 12 years of follow-up (patients are followed up to 13 years).
OS in SER patients | Time from randomization to death due to any cause, assessed up to 12 years after the last enrollment
  Will be compared between a standard chemotherapy approach and an IO therapy approach among the SER patients.
OS for entire patient population | Time from randomization to death due to any cause, assessed at 12 years after the last enrollment
  Will be based on a confidence interval approach conducted after the last patient not lost to follow-up has been followed for at least 12 years from randomization. Twelve-year OS and its corresponding 90% confidence interval will be estimated with the Kaplan-Meier method for each study arm within the entire randomized and evaluable trial population.
PFS for favorable risk patients | Up to 12 years
  Will be estimated in patients with favorable features at diagnosis. PFS and a corresponding confidence interval will be estimated using the Kaplan-Meier approach. PFS will also be compared between the (pooled) IO therapy and standard therapy arms using stratified log-rank tests within each cohort.
PFS for unfavorable risk patients | Up to 12 years
  Will be estimated in patients with unfavorable features at diagnosis. PFS and a corresponding confidence interval will be estimated using the Kaplan-Meier approach. PFS will also be compared between the (pooled) IO therapy and standard therapy arms using stratified log-rank tests within each cohort.
PFS for entire population | Up to 12 years
  PFS and a corresponding confidence interval will be estimated using the Kaplan-Meier approach. PFS will also be compared between the (pooled) IO therapy and standard therapy arms using stratified log-rank tests within each cohort.
Event-free survival (EFS) | Time from randomization to the earliest of progression, relapse, second malignancy, or death due to any cause, assessed up to 12 years from last enrollment
  Pooling IO treatment arms and standard treatment arms, EFS and corresponding confidence intervals will be estimated with the Kaplan-Meier approach for patients assigned versus (vs.) not assigned to receive radiaton therapy (RT), and compared using the log-rank test.
Incidence of adverse events (AEs) | Assessed up to 12 years from last enrollment
  Will use the American Society of Clinical Oncology and the Society for Immunotherapy of Cancer guidelines to capture immune-related AEs. Physician-reported treatment related AEs will be reported for all grades using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Rates of individual toxicities with grades greater or equal to 3 will be compared between the pooled IO and standard arms using exact binomial tests. The maximum grade for each toxicity will be recorded for each patient. The rates and confidence intervals for these toxicities will be provided. Comparison of AEs will also be conducted for physician-reported treatment-related AEs between RT and non-RT patients.
Patient reported outcomes (PRO)-CTCAE | Assessed up to 12 years from last enrollment
  Targeted patient-reported AEs will be collected at each time point using the PRO-CTCAE for patients 7 years and older. For youth (7-17 years) the Pediatric PRO-CTCAE form will be used and for those 18 years and older adult the PRO-CTCAE form will be used. For information collected by each of the above forms, the scores for each attribute together with frequency, severity and/or interference will be presented descriptively using summary statistics at each assessment time. Additionally, the worst severity and/or interference over the entire course will be summarized. The changes among main time points will be calculated. The results will be provided for the whole population and compared between subpopulations by arms and by age groups. Regression models based on longitudinal measurements can be constructed by considering the following covariates besides age groups: baseline demographics, clinical risk factors, and study arms.
Patient-reported fatigue | Baseline up to 1 year from end of study treatment
  Will be measured by validated short forms from the Patient Reported Outcomes Measurement Information System initiatives. Domain scores will be converted to T-scores with an established standard deviation of 10 points with an average score normalized to 50 within the healthy adult population. The minimal clinically important difference (MCID) in these PRO measures has been accepted to be 2-3 points of the standard deviation (SD = 10) of the measure. To account for the dual primary PRO outcomes of fatigue and cognitive deficits, we will consider Bonferroni correction of p-values. Primary interests will be differences in T-scores between IO and chemotherapy arms at 1-year post completion of therapy.
Patient-reported cognitive deficits | Baseline up to 1 year from end of study treatment
  Will be measured by validated short forms from the Neuro-QoL initiative. Domain scores will be converted to T-scores with an established standard deviation of 10 points with an average score normalized to 50 within the healthy adult population. The MCID in these PRO measures has been accepted to be 2-3 points of the standard deviation (SD = 10) of the measure. To account for the dual primary PRO outcomes of fatigue and cognitive deficits, we will consider Bonferroni correction of p-values. Primary interests will be differences in T-scores between IO and chemotherapy arms at 1-year post completion of therapy.
Patient-reported health-related quality of life | Baseline up to 1 year from end of study treatment
  Domain scores will be converted to T-scores with an established standard deviation of 10 points with an average score normalized to 50 within the healthy adult population. The MCID in these PRO measures has been accepted to be 2-3 points of the standard deviation (SD = 10) of the measure. To account for the dual primary PRO outcomes of fatigue and cognitive deficits, we will consider Bonferroni correction of p-values. Primary interests will be differences in T-scores between IO and chemotherapy arms at 1-year post completion of therapy.
Incidence of self-reported late morbidities | Assessed up to 12 years from last enrollment
  Will be collected by using validated measures from the St. Jude Life Cohort. The cumulative incidence of late-morbidities (e.g., cardiovascular, pulmonary and endocrine) will be compared between the standard chemotherapy and the IO therapy and among different age groups (7-14; 15-40 and 41-60) with K-sample method. The frequencies of selected organ toxicities will be compared between two treatment arms, among the three age groups and between RT and non-RT with chi-square tests.
Effect of metabolic tumor burden (MTV) on PFS | At baseline prior to initiation of therapy
  MTV will be measured at baseline using fludeoxyglucose F-18 (FDG)-PET. The Kaplan-Meier curves of PFS will be compared between the two levels with log-rank tests.
Effect of total lesion glycolysis (TLG) on PFS | At baseline prior to initiation of therapy
  TLG will be measured at baseline using FDG-PET. The Kaplan-Meier curves of PFS will be compared between the two levels with log-rank tests.
Contribution of social determinants of health (SDOH) to PET2 response by race and ethnicity | After Cycle 2 of treatment (1 cycle = 28 days)
Contribution of SDOH to PFS by race and ethnicity | Assessed up to 12 years after last enrollment
  Kaplan-Meier (K-M) curves of PFS will be generated by racial/ethnic groups (e.g., non-Hispanic white [NHW], non-Hispanic black [NHB], Hispanic). The p values for the K-M curve comparison will be obtained from log-rank tests. Associations between race/ethnicity and PFS will be evaluated with univariable and multivariable Cox proportional hazard models by considering other covariates such as baseline clinical conditions, toxicities, SDOH, and treatment arm (standard vs. IO). Backward selection will be used to select those factors with p-value < 0.2, which will be included in final multivariable models.
Contribution of SDOH to OS by race and ethnicity | Assessed up to 12 years after last enrollment
  K-M curves of OS will be generated by racial/ethnic groups (e.g., NHW, NHB, Hispanic). The p values for the K-M curve comparison will be obtained from log-rank tests. Associations between race/ethnicity and OS will be evaluated with univariable and multivariable Cox proportional hazard models by considering other covariates such as baseline clinical conditions, toxicities, SDOH, and treatment arm (standard vs. IO). Backward selection will be used to select those factors with p-value < 0.2, which will be included in final multivariable models.

OTHER OUTCOMES:
PFS comparison between treatment arms for each age group | Up to 12 years
  Will be compared between a standard chemotherapy approach and an IO therapy approach within different age groups (ages 5-11 years, 12-21 years, 22-39 years, 40-60 years) using log-rank tests. Cox regression models will be constructed to evaluate the treatment effects for different age groups while considering the impact of other potentially prognostic variables including baseline demographics and clinical risk factors. PFS and corresponding confidence intervals for each age group will be estimated with the Kaplan-Meier method, overall and by treatment arms. In additional models, age may be evaluated as a continuous variable with potentially non-linear effects on PFS.
Concordance and discordance of 5-point score (PS) visual PET assessments | At baseline, post cycle 2, and at end of systemic therapy
  The concordance and discordance of 5-PS visual PET assessment from rapid central review and local institutional review will be evaluated at each of the timepoints. Will collect and retrospectively review local vs. central review concordance rates. For discordant cases, will document the differences in treatments if only local review or only central review were performed
Association between FDG PET parameters obtained by automated measurements and PFS | At baseline, post cycle 2, and at the end of therapy
  The association between FDG PET parameters obtained by automated measurements using convolutional neural networks and PFS will be evaluated in this aim. The PET parameters of interest are total MTV and TLG, tumor standardized uptake value change. PET parameters will be obtained based on artificial intelligence (AI) based measurements. The effect of these PET measurements will be evaluated by Cox regression models.
Agreement between AI derived FDG-PET measurement extraction and physician-based manual quantitative PET measurement | At baseline, post cycle 2, and at the end of therapy
  Will compare AI derived automated quantitative FDG-PET measurement extraction and physician-based manual quantitative PET measurement with Spearman rank correlation coefficients for each extracted PET metric.
Incidence of patient reported adverse events and provider adverse event reporting | Assessed up to 12 years
  Will be collected by PRO-CTCAE and Ped-PRO-CTCAE. The patient reported AEs will be compared to provider reported AEs reported descriptively.
Association between self-reported race/ethnicity and dimensional SDOH | Assessed up to 12 years
  Will be evaluated by Chi-square tests or Fisher exact tests for sparse data. Will also calculate the area deprivation index (derived from patient-reported address and zip code to census block-group data for patients treated in the United States, and the Canadian Index of Multiple Deprivation for patients treated in Canada) and investigate its association with race/ethnicity and SDOH.
Post-relapse/post-progression OS by race/ethnicity and select SDOH measures | Assessed up to 12 years
  The K-M curves will be presented together with p-values via log-rank tests across the different race/ethnicity groups for each treatment arm. Cox proportional hazard models to evaluate the relationship between race/ethnicity and post-relapse OS will be constructed.
Completion rate of PRO and health-related quality of life contact forms | At 1 year off treatment
  Will be evaluated for the first 450 eligible participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kara M Kelly, Principal Investigator — Roswell Park Cancer Institute
Locations (395):
- United States (380):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Corona, Corona, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - City of Hope Seacliff, Huntington Beach, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - City of Hope Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794